CLINICAL TRIAL: NCT07053046
Title: PRECIDENTD Engagement Methods for Sites (PRECIDENTD-EMS)
Brief Title: PRECIDENTD Engagement Methods for Sites
Acronym: PRECIDENTD-EMS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lyndsay Nelson, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 250764; SOE-2024C1-37523 (Other Grant/Funding Number: PCORI)
Record Dates: First submitted 2025-06-30; First posted 2025-07-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Stakeholder Engagement
Keywords: Stakeholders; Engagement; Agile Methods; Patient Partners

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard engagement approach (Placebo Comparator)
  Interventions: Other: Standard engagement approach
- Agile methods engagement approach (Experimental)
  Interventions: Other: Agile methods engagement approach

INTERVENTIONS:
Other: Standard engagement approach — Large group meetings led by PRECIDENTD PIs; composed of ~20 sites (with ~25 site investigators and ~40 study staff). PRECIDENTD PIs will share updates and facilitate discussion around any problems.
  Problem identification and steps toward solution occur sequentially. A problem is identified in the data (e.g., slow recruitment), then brought to the Stakeholder Advisory Council (SAC) for advisement, then back to site investigators and study staff to implement recommended changes, the PIs look at data to see if changes improved the problem. PIs and the Stakeholder Engagement Core broker information and relationships with SAC partners.
  Arms: Standard engagement approach
Other: Agile methods engagement approach — Small group meetings led by a coordinator trained in agile methods; composed of ~4 sites each (representing 4-6 investigators and 6-10 study staff), plus 2-3 Stakeholder Advisory Council (SAC) patient partners. Meetings will focus on problem-solving around specific topics and apply agile tools and principles.
  Sites in each small group will review process data together and each site will identify a specific topic (recruitment, retention, medication adherence) to focus on improving over the next month. Research partners at sites and patient partners will contribute to discussion and reflection on barriers, challenges, successes, and facilitators. Steps toward solutions occur on a rapid timeframe, iteratively using data as a guidepost.
  Arms: Agile methods engagement approach

SUMMARY:
This trial is evaluating approaches to effective stakeholder engagement as part of an ongoing multi-site trial, called PRECIDENTD (PREvention of Cardiovascular and DiabEtic kidNey disease in Type 2 Diabetes). PRECIDENTD is a PCORI-funded trial comparing two classes of medication for reducing major health events (e.g., heart attack, stroke, kidney disease) in patients with type 2 diabetes. This is a trial within PRECIDENTD examining Engagement Methods for Sites (PRECIDENTD-EMS) in which PRECIDENTD study sites are randomized to agile engagement methods or a standard engagement approach. The application of agile methods will provide opportunities for increased collaboration between patient partners and study sites during the conduct of the study. The hypothesis is that this will result in better research outcomes for the larger PRECIDENTD study, as well as engagement quality and partner outcomes among those engaged with the conduct of the PRECIDENTD study, as compared with a standard engagement approach.

This study is designed to assess if agile methodology - when applied to engagement during the conduct of a study - will affect research outcomes of that study, as well as the quality of engagement.

Aim 1: Evaluate whether agile methods applied to stakeholder engagement impact research outcomes. The investigators will compare research outcomes (recruitment, adherence to assigned medication, and retention in the larger PRECIDENTD study) between study sites in the agile and standard engagement arms.

Aim 2. Evaluate whether agile methods in stakeholder engagement impact partners and identify potential mediators of effects. The investigators will examine engagement quality and partner outcomes between the agile and standard engagement arms. The investigators will also explore engagement quality as a potential driver/mediator of the effects of agile methods on partner outcomes.

ELIGIBILITY:
Inclusion Criteria:

* PRECIDENTD patient stakeholder advisory council partners
* PRECIDENTD site study staff
* PRECIDENTD site investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Participant Recruitment | 18 months post-baseline
  Total patient participants enrolled in PRECIDENTD across sites
Engagement experience | Baseline and 6, 12, and 18 months post-baseline
  As measured by the Patient Engagement in Research Scale (PEIRS); Procedural requirements and Convenience subscales. Items scored on a scale from 0-5, where higher scores indicate better engagement experiences.
Partnership functioning | Baseline and 6, 12, and 18 months post-baseline
  As measured by the Patient Engagement in Research Scale (PEIRS); Contributions and Support subscales. Items scored on a scale from 0-5, where higher scores indicate better partnership functioning.
Group dynamics | Baseline and 6, 12, and 18 months post-baseline
  As measured by the Patient Engagement in Research Scale (PEIRS); Team environment and interaction subscale. Items scored on a scale from 0-5, where higher scores indicate better group dynamics.
Equity and Inclusiveness | Baseline and 6, 12, and 18 months post-baseline
  Selected & adapted items from the Research Engagement Survey Tool (REST) - Facilitate collaborative, equitable partnerships subscale. Items scored on a scale from 0-5, where higher scores indicate better equity and inclusiveness.

SECONDARY OUTCOMES:
Medication adherence | Baseline and 18 months
  Proportion of PRECIDENTD study participants taking assigned study medication across sites. As assessed by participant self-report via communication with study sites and study assessments.
Participant retention | Baseline and 18 months
  Proportion of PRECIDENTD study participants completing study visits across sites.
Participant retention | Baseline and 18 months
  Proportion of PRECIDENTD study participants completing study assessments across sites.
Post-engagement capacity and readiness | 12 and 18 months post-baseline
  Item developed by the study team. Items scored on a scale from 0-5, where higher scores indicate better post-engagement capacity and readiness.
Costs and benefits | Baseline and 6, 12, and 18 months post-baseline
  Selected & adapted items from the Patient Engagement in Research Scale (PEIRS); Benefits subscale. Items scored on a scale from 0-5, where higher scores indicate better benefits.
Engagement Sustainability | 12 and 18 months post-baseline
  Selected & adapted items from the REST - Partnership sustainability to meet goals and objectives. Items scored on a scale from 0-5, where higher scores indicate better engagement sustainability.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to share IPD data, but have not yet developed a specific plan.